CLINICAL TRIAL: NCT00823342
Title: ANRS HB 05 : A Randomized, Double Blind, Multicenter Study Evaluating Efficacy and Safety of Clevudine Monotherapy Versus Tenofovir Monotherapy Versus Combination Therapy of Clevudine and Tenofovir for 96 Weeks in HBeAg Negative Patients With Chronic Hepatitis B, naïve to Anti-VHB Therapy
Brief Title: ANRS HB 05 Multicenter Study Evaluating Efficacy and Safety of Clevudine Monotherapy Versus Tenofovir Monotherapy Versus Combination Therapy of Clevudine and Tenofovir for 96 Weeks in HBeAg Negative Patients With Chronic Hepatitis B, naïve to Anti-VHB Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: safety aspects
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Gilead Sciences (Industry); Pharmasset (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-000733-21; ANRS HB 05
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: HBe Negative Chronic Hepatitis B; Hepatitis B Viral Infection
Keywords: HBe, Hepatitis, Vireda (TENOFOVIR, CLEVUDINE), HBV, HBe Ag negative
MeSH Terms: conditions — Hepatitis; Hepatitis B | interventions — clevudine; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Placebo Comparator): CLEVUDINE 30 mg qd + TENOFOVIR Placebo
  Interventions: Drug: CLEVUDINE + TENOFOVIR PLACEBO
- Group B (Active Comparator): TENOFOVIR 300 mg qd in association with CLEVUDINE 30 mg qd
  Interventions: Drug: CLEVUDINE IN ASSOCIATION TENOFOVIR
- Group C (Placebo Comparator): TENOFOVIR 300 mg qd + CLEVUDINE Placebo
  Interventions: Drug: TENOFOVIR + CLEVUDINE PLACEBO

INTERVENTIONS:
Drug: CLEVUDINE + TENOFOVIR PLACEBO — 30 MG
  Arms: Group A
Drug: CLEVUDINE IN ASSOCIATION TENOFOVIR — TENOFOVIR 300 mg qd in association with CLEVUDINE 30 mg qd
  Arms: Group B
Drug: TENOFOVIR + CLEVUDINE PLACEBO — TENOFOVIR 300 mg qd + CLEVUDINE Placebo
  Arms: Group C

SUMMARY:
For chronic HBV infection, an optimal pharmacological agent to promote recovery from chronic HBV infection would be one that inhibits HBV DNA polymerase, combined with the clearence from the liver of cccDNA to block HBV reactivation after the circulating viral burden has been eliminated by therapy. The activity of clevudine on cccDNA in combination with its potent antiviral activity on HBV polymerase makes it the optimal agent in combination with tenofovir for this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over 18 years of age
* Chronic hepatitis B, HBs Ag-positive for over 6 months, anti HBs negative
* Patients with HBeAg- negative chronic hepatitis B (CHB) and anti-HBe positive at screen
* Patients naïve to anti-HBV nucleoside or nucleotide and any other experimental nucleoside/nucleotide analog for HBV
* Serum HBV-DNA quantifiable over 2000 IU/mL at screening
* ALT over 1.25 ULN and below 10 ULN
* Liver biopsy (baseline or within prior 6 months) with evidence of chronic hepatic inflammatory injury (Metavir Activity score over 1 ; Knodell necroinflammatory score over 3, Ishak score over 1)

Exclusion Criteria:

* Cirrhosis or bridging fibrosis on liver biopsy
* Subjects who have received any form of alpha interferon in the past 6 months prior to the first administration of randomized treatment
* Any systemic anti-viral, anti-neoplastic or immuno-modulatory treatment (including supraphysiologic doses of steroids and radiation) below 6 months prior to the first dose of randomized treatment and during the study (except for below 10 days of acyclovir for herpetic lesions, or prednisone below 10 mg/days for below 10 days more than 1 month)
* Women with ongoing pregnancy or breast feeding
* Positive test at screening for anti-HAV IgM Ab, anti-HIV Ab, anti-HCV Ab, HCV RNA, anti-HDV Ab
* History or other evidence of a medical condition associated with chronic liver disease other than HBV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease including Wilson's disease and alpha1-antitrypsin deficiency, alcoholic liver disease, toxin exposures, toxic thalassemia, NASH)
* History or other evidence of bleeding from esophageal varices or other clinical conditions consistent with decompensated liver disease (defined by one of the following criteria being met: serum albumin below 3.5 g/L, prothrombin time over 4 seconds prolonged, serum bilirubin over 34 µmol/L, history of encephalopathy, history of ascites)
* Neutrophil count below 1200 cells/mm3 or platelet count below 90,000 cells/mm3 at screening
* Serum creatinine level over 130µmol/l or calculated creatinine clearance below 70 ml/min (Cockcroft-Gault)
* Evidence or history of tubular nephropathy , Fanconi syndrom or hypophosphoremia.
* Evidence of drug abuse (including excessive alcohol consumption) within one year of study entry
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis etc.)
* History of major organ transplantation with an existing functional graft
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Evidence of an active or suspected cancer or a history of malignancy where the risk of recurrence is over 20 % within 2 years
* Patients with a value of alpha-fetoprotein over 100 ng/mL are excluded, unless stability (less than 10 % increase) has been documented over at least the previous 3 months
* Patients included in another trial within 8 weeks prior to screening
* Inability or unwillingness to provide informed consent or abide by the requirements of the study Reassessments : If a patient fails to meet the above inclusion /exclusion criteria for a reason thought to be reversible, that patient may be reassessed for entry on two additional occasions at most. If the parameter out of range for inclusion was ALT over 10 x ULN, the patient should be reassessed over 4 weeks after the date corresponding to the value that was over 10 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-12-14 (Actual); Primary Completion 2008-12-14 (Actual); Study Completion 2008-12-14 (Actual)

PRIMARY OUTCOMES:
Compare the long term efficacy of new anti-HBV strategies of CLV monotherapy VS TDF monotherapy VS the combination of CLV + TDF for 96 weeks in HBeAg negative patients with CHB, naïve to anti-HBV-therapy, at 24 weeks post-treatment | At 120 week

SECONDARY OUTCOMES:
Compare the safety profile of CLV + TDF compared to that of CLV and TDF in HBeAg negative patients with CHB, naïve to anti-HBV-therapy. - To compare perceived toxicity as expressed by the nature and the number of self-reported side effects, percept | At 24 week, 48 week and 96 week

CONTACTS AND LOCATIONS:
Overall Officials: MARC BOURLIERE, MD, Principal Investigator — Hôpital Saint Joseph, marseille, France
Locations (1):
- Hôpital Saint Joseph, Marseille, France